CLINICAL TRIAL: NCT07141498
Title: Evaluation of i-Gel and Air-Q sp3G Supraglottic Airway Device Placement by Fiberoptic Bronchoscopy and Comparison of Gastric Insufflation Volumes Using Ultrasound in Pediatric Patient
Brief Title: Fiberoptic Evaluation of i-Gel and Air-Q sp3G Supraglottic Airway Devices in Pediatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: igelvsAirqFOB
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Laryngeal Mask Airways; Fiberoptic Bronchoscopy (FOB); Elective Surgeries; Gastric Insufflation; Gastric Ultrasound
Keywords: laryngeal mask; airway management; ultrasonography; child

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- igel: Pediatric patients aged 1-8 years undergoing elective pediatric or urological surgery under general anesthesia. Supraglottic airway (SGA) management will be performed using the igel second-generation device. Position verification will be performed via fiberoptic bronchoscopy (Grade 3-4 accepted as correct). Gastric volume will be measured with USG pre-insertion, post-insertion, and at surgery completion. Pre-, intra-, and postoperative complications will be documented as in the iGel group.
- Air-Q sp3G: Pediatric patients aged 1-8 years undergoing elective pediatric or urological surgery under general anesthesia. Supraglottic airway (SGA) management will be performed using the Air-Q sp3G second-generation device. Position verification will be performed via fiberoptic bronchoscopy (Grade 3-4 accepted as correct). Gastric volume will be measured with USG pre-insertion, post-insertion, and at surgery completion. Pre-, intra-, and postoperative complications will be documented as in the iGel group.

SUMMARY:
This single-center, prospective, randomized controlled study aims to compare the placement accuracy of iGel and Air-Q sp3G supraglottic airway (SGA) devices in pediatric patients aged 1-8 years undergoing elective surgery under general anesthesia. Placement will be confirmed via fiberoptic bronchoscopy, and gastric insufflation will be assessed using ultrasound measurement of gastric antral cross-sectional area pre- and post-device placement. Secondary outcomes include postoperative complications such as sore throat, hoarseness and dysphagia.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled trial will be conducted in pediatric patients aged 1-8 years undergoing elective pediatric or urological surgery under general anesthesia. Participants will be randomized into two groups to receive either an iGel or an Air-Q sp3G device. Device placement will be confirmed intraoperatively via fiberoptic bronchoscopy using a standardized grading system and gastric antral cross-sectional area will be measured with ultrasound before device insertion, immediately after insertion and at the end of surgery to evaluate gastric insufflation.

Secondary outcomes will include postoperative complications such as sore throat, hoarseness, dysphagia, mucosal bleeding, cough, laryngospasm, bronchospasm, nausea, vomiting and stridor. Intraoperative variables such as number of insertion attempts, ease of placement and peak airway pressure will also be recorded. The results are expected to identify which device offers better placement accuracy and lower gastric insufflation rates, thereby improving perioperative safety and postoperative recovery in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-8 years
* ASA I-III
* Elective pediatric or urological surgery under general anesthesia with SGA use
* Informed consent obtained from parents/guardians

Exclusion Criteria:

* Parental refusal or inability to consent
* ASA > III
* Recent or current upper respiratory tract infection
* History of difficult airway
* Increased aspiration risk
* Urgent/emergency surgery or non-fasted patients
* Known allergy or contraindication to anesthetic agents
* Severe asthma (attack within last 6 months)
* Structural airway anomalies
* Gastrointestinal pathology affecting stomach emptying
* Previous stomach surgery

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 1-8 years (ASA I-III) undergoing elective pediatric surgery under general anesthesia at Ankara Bilkent City Hospital. Eligible participants will require supraglottic airway device placement (i-Gel or Air-Q sp3G).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Correct SGA Placement Rate via Fiberoptic Bronchoscopy | Device placement will be assessed intraoperatively
  In pediatric patients undergoing elective surgery under general anesthesia, the correct placement of supraglottic airway devices (iGel vs. Air-Q sp3G) will be assessed using fiberoptic bronchoscopy grading (Grade 3-4 considered correct positioning).
Gastric insufflation volume | gastric volume will be measured intraoperatively
  Gastric volume will be measured by ultrasound (USG) at three time points:
  Baseline (pre-induction): After IV induction, in supine position, before SGA insertion.
  Post-SGA insertion: Immediately after supraglottic airway (i-Gel or Air-Q sp3G) placement.
  End of surgery: Before emergence from anesthesia. The change in gastric volume across these time points will be compared between i-Gel and Air-Q sp3G groups.

SECONDARY OUTCOMES:
Peak Airway Pressure | Intraoperative - immediately after insertion
  Peak inspiratory airway pressure measured intraoperatively after SGA placement
Number of Attempts for Successful SGA Placement | Intraoperative
  Count of insertion attempts required to achieve correct SGA positioning
Postoperative Sore Throat | 6 hours postoperative
  Incidence of sore throat assessed by direct questioning at 6 hours after surgery.
Postoperative Hoarseness | 6 hours postoperative
  Incidence of hoarseness assessed by direct questioning at 6 hours after surgery.
Postoperative Dysphagia | 6 hours postoperative
  Incidence of swallowing difficulty assessed at 6 hours after surgery
Incidence of mucosal bleeding | 6 hours postoperative
  Incidence of mucosal bleeding assessed by direct questioning at 6 hours after surgery.
Incidence of nausea | 6 hours postoperative
  Incidence of nausea assessed by direct questioning at 6 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Department Of Anesthesiology and Reanimation, Ankara, Turkey (Türkiye)